CLINICAL TRIAL: NCT00647595
Title: Effect of Physical Activity on Metabolic Syndrome in Pregnancy & Fetal Outcome
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Lee, Sum P MD, Phd, Professor of Medicine, University of Washington School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: R03 DK74683 (completed); NIH # 1 R03 DK074683-01A1; R03DK074683 (NIH)
Record Dates: First submitted 2008-03-27; First posted 2008-03-31 (Estimated); Last update posted 2015-04-22 (Estimated); Status verified 2010-02

CONDITIONS: Obesity; Pregnancy; Diabetes Mellitus
Keywords: Obesity; Physical activity; Pregnancy; Diabetes mellitus
MeSH Terms: conditions — Obesity; Diabetes Mellitus; Motor Activity

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Experimental): Women in this group will exercise 3x per week at a moderate/vigorous level for 45 min per session through their 36 week of pregnancy.
  Interventions: Behavioral: Experimental group
- B (No Intervention): Women in this group will continue their usual activities throughout their pregnancy.

INTERVENTIONS:
Behavioral: Experimental group — Intervention group will exercise 3 times per week at moderate-vigorous intensity for 45 minutes per session. Control group women will continue their usual physical activity throughout pregnancy.
  Arms: A

SUMMARY:
The purpose of this study is to examine the effect of exercise during pregnancy upon maternal metabolism, including weight gain, fat distribution, and levels of glucose and cholesterol. We will also conduct a pilot study to examine the feasibility of studying the health of infants born to women in this study.

DETAILED DESCRIPTION:
Obesity and overweight have become important public health problems in the United States, and measures are urgently needed to address these issues. For many women, pregnancy is a time of excessive weight gain and decreases in physical fitness, both of which may be followed by postpartum weight retention. Women who develop hypertension or diabetes mellitus during pregnancy are at higher risk for development of these disorders in the future. Because of the implications of pregnancy-related weight gain and the metabolic changes during pregnancy for future maternal health, interventions to maintain or improve fitness during pregnancy may have important downstream health effects. In addition, maternal metabolic parameters and the intra-uterine environment have important implications for neonatal outcomes and subsequent child health. This study will provide data about the effects of an intervention to increase vigorous physical activity during pregnancy on short-term maternal and fetal outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women 18-45 years old receiving prenatal care at MAMC

Exclusion Criteria:

* Women do not have a gallbladder
* Who do not speak English
* Are over 14 weeks pregnant at study entry
* Do not plan to deliver at MAMC
* Have medical contraindications
* Unwilling to participate in exercise intervention program
* Are under 18 years of age
* Currently engaged in a regular vigorous exercise program

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2007-10; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Central adiposity | 6-8 weeks postpartum

SECONDARY OUTCOMES:
Leptin levels | during pregnancy and postpartum
glucose | during pregnancy and postpartum
insulin | during pregnancy and postpartum
cholesterol | during pregnancy and postpartum
fetal adiposity | 35-36 weeks gestation
neonatal adiposity | birth

CONTACTS AND LOCATIONS:
Overall Officials: Cynthia W Ko, MD MS, Principal Investigator — University of Washington
Locations (1):
- Madigan Army Medical Center, Joint Base Lewis McChord, Washington, United States